CLINICAL TRIAL: NCT02661620
Title: A Retrospective-Prospective Study of REDAPT™ Revision Femoral System Modular Stem
Brief Title: REDAPT Retrospective-Prospective Modular Stem Study
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely terminated by S+N due to business reasons. After an extensive review of all ongoing studies with the focus on which studies are still required for regulatory obligations S+N took the decision to close the REDAPT 15 study.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REDAPT 15-4538-02
Record Dates: First submitted 2016-01-12; First posted 2016-01-22 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Arthroplasties, Hip Replacement
Keywords: REDAPT Femoral System modular stem implant; Total Hip arthroplasty revision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: REDAPT Revision Femoral System modular stem — Medical record review for retrospective information and observational prospective data collection of standard of care items at 5 years and 10 years post operatively plus a 7.5 year post op telephone call to assess stem status and adverse events.

SUMMARY:
A Retrospective-Prospective Study of REDAPT Revision Femoral System Modular Stem is a post-market, retrospective-prospective, multi-center, single arm, consecutive series study design to provide data on the post market performance and safety of the study device. The study will collect retrospective data from medical records review and prospective data from observations data at 5 and 10 postoperatively clinical visits. There will also be a 7.5 year telephone follow up contact to assess for device status and adverse events.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate the REDAPT™ Revision Femoral System modular stem cumulative revision rate at 5 years.

The secondary purpose of this study is to provide 10 years of safety and performance data on the REDAPT™ Revision Femoral System modular stem in terms of Standard of Care Radiographic Assessment, Harris Hip Sore (if obtained prior to implant), adverse event assessment, whole blood metal ion level assessment for Cobalt and Chromium (only performed if subject if symptomatic with pain, swelling, and/or functional limitation related to the device and/ implant procedure as assessed by the Principal Investigator (PI), and Metal artifact reduction sequence (MARS) magnetic resonance imaging (MRI) or Computed Tomography (CT) will be obtained if metal ion levels of Cobalt and/or Chromium > 7parts per billion (ppb) 140 subjects have been enrolled in the study at 5 clinical study sites around the world. A Clinical Study Report (CSR) will be completed at years 5 and 10.

ELIGIBILITY:
Inclusion Criteria:

Retrospective Limited Data Collection/Enrollment Phase:

• Subject has undergone revision hip arthroplasty with the REDAPT™ Revision Femoral System modular stem with implantation from 2012 to the date of Institutional Review Board (IRB)/Ethics Committee (EC) approval ofthe original version 1.0 protocol at the study site.

Retrospective Expanded Data Collection & Prospective Follow-Up Phase:

* Subject completed limited retrospective data collection phase and willing to consent to expanded retrospective data collection and the prospective phase of the study;
* Subject is willing and able to participate in required follow-up visits at the investigational site and to complete study procedures.

Exclusion Criteria:Retrospective Limited Data Collection/Enrollment Phase:

• Not applicable

Retrospective Expanded Data Collection & Prospective Follow-Up Phase:

* Subject, in the opinion of the PI, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse; or
* Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject has undergone revision hip arthroplasty with the REDAPT™ Revision Femoral System modular stem with implantation from 2012 to the date of Institutional Review Board (IRB)/Ethics Committee (EC) approval of this protocol at the study site.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Modular stem revision | 5 years post operatively
  Listing of stem implant status at 5 years to analyze stem survival rate

SECONDARY OUTCOMES:
Revision of any component for any reason | 5 year post operative
  revision for any reason
Radiographic assessments | follow-up to 10 years as per standard of care
  radiographic measurements to assess linear radiolucencies and subsidence to assess safety and potential changeover time
Harris Hip Score | collect retrospectively from medical record preoperative and if done preoperatively at 1 year, 5 year and 10 year follow up visits
  Clinical evaluation to score and assess changes over time from baseline through 10 year post.
Adverse Events | through study completion, an average of 10 years
  Adverse events will be collected to monitor the safety, retrospectively from medical record review starting with operative date through end of study

OTHER OUTCOMES:
Whole blood metal ion level assessment for cobalt and chromium | through study completion, an average of 10 years
  performed for subject if symptomatic with pain, swelling, and/or functional limitation related to the device and/ implant procedure as assessed by the Principal Investigator (PI)
MARS MRI or CT images acquired pending outcome of whole blood metal ion level assessment | based on results of outcome 6, through study completion, an average of 10 years
  Metal artifact reduction sequence (MARS) magnetic resonance imaging (MRI) or Computed Tomography (CT) will be obtained if metal ion levels of Cobalt and/or Chromium > 7parts per billion (ppb)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jahnke, Study Chair — Smith & Nephew, Inc.
Locations (5):
- United States (3):
  - Baptist Health Louisville Orthopedic, Louisville, Kentucky
  - Detroit Receiving Hospital, Detroit, Michigan
  - The Oregon Health & Science University, Portland, Oregon
- ZNA Campus Middelheim, Antwerpe, Antwerp, Belgium
- CHU De Quebec- Hôpital Saint-François d'Assise, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No